CLINICAL TRIAL: NCT00040677
Title: A Phase II, Multicenter, Twelve-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Range-Finding Study of the Efficacy and Safety of ICA-17043 With or Without Hydroxyurea Therapy in Patients With Sickle Cell Anemia
Brief Title: A Study of the Efficacy and Safety of ICA-17043 (With or Without Hydroxyurea) in Patients With Sickle Cell Anemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icagen (Industry)
Responsible Party: Greg Rigdon, Vice President New Product Development, Icagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICA-17043-05
Record Dates: First submitted 2002-07-08; First posted 2002-07-10 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: sickle cell anemia; sickle cell disease; anemia; ICA-17043; senicapoc
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — senicapoc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ICA-17043 Low Dose 6 mg/day (Experimental): Active study medication: 100 mg loading dose; 6 mg maintenance dose per day
  Interventions: Drug: Low Dose ICA-17043
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ICA-17043 High Dose 10 mg/day (Experimental): Active study medication: 150 mg loading dose; 10 mg maintenance dose per day
  Interventions: Drug: High dose ICA-17043

INTERVENTIONS:
Drug: Low Dose ICA-17043 — Low dose arm
  Arms: ICA-17043 Low Dose 6 mg/day
Drug: High dose ICA-17043 — 150 mg Loading Dose; 10 mg daily dose
  Arms: ICA-17043 High Dose 10 mg/day
Drug: Placebo — Placebo Loading dose capsules and maintenance dose tablets matched 10 mg active treatment group
  Arms: Placebo

SUMMARY:
ICA-17043 is being developed for the chronic treatment of patients with sickle cell disease (SCD) in both adults and children. ICA-17043 is a potent and specific inhibitor of a channel in human red blood cells (RBCs) that blocks RBC dehydration. ICA-17043 is expected to inhibit RBC dehydration and thus should prevent or delay the sickling process. By reducing sickled cells, an improvement in anemia, a reduction in painful crises, and ultimately, less end-organ disease is anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous (HbSS) Sickle Cell Anemia
* Otherwise healthy (based on medical history, physical examination, 12-lead ECG, and clinical laboratory tests)
* Patients may be receiving hydroxyurea, but must have been dose stabilized for at least 3 months
* Patient has a history of at least one acute vaso-occlusive event requiring hospitalization

Exclusion Criteria:

* Patient participating in a chronic transfusion program
* Patient having a total hemoglobin of < 4.0 g/dL or > 10.0 g/dL
* Patient having a HbA > 10%
* Patient considering undergoing an elective surgery
* Patient taking prohibited medications such as Epoetin, Warfarin, etc.
* Patient who has had previous gastrointestinal surgery, except cholecystectomy or appendectomy
* Patient with significant active cardiovascular, neurologic, endocrine, hepatic, or renal disorders unrelated to sickle cell anemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2002-02; Primary Completion 2003-11 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the change from Baseline in hemoglobin (Hb) | 12 Weeks

SECONDARY OUTCOMES:
Changes in other hematologic measurements | 12 weeks
Changes in RBC indices, including: mean corpuscular volume (MCV), mean corpuscular Hb concentration (MCHC), and mean corpuscular Hb (MCH | 12 weeks
Other laboratory measures associated with sickle cell crises activity including: direct and indirect bilirubin and lactic dehydrogenase (LDH) | 12 weeks
Rate of painful crises | 12 weeks
Time to first painful crisis | 12 weeks
Morbidity of painful crises (maximum morbidity index, derived variable) | 12 weeks
Pain intensity scores | 12 weeks
Quality of Life (SF 36) | 12 Weeks
Health economic data | 12 weeks
Average plasma concentration | 12 weeks
Correlation between the average plasma concentration and the change in Hb from Baseline to study endpoint | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (19):
- United States (19):
  - Study Site, Birmingham, Alabama
  - Study Site, Oakland, California
  - Study Site, San Francisco, California
  - Study Site, Washington D.C., District of Columbia
  - Study Site, Augusta, Georgia
  - Study Site, Chicago, Illinois
  - Study Site, Baltimore, Maryland
  - Study Site, Boston, Massachusetts
  - Study Site, Detroit, Michigan
  - Study Site, Jackson, Mississippi
  - Study Site, Brooklyn, New York
  - Study Site, New York, New York
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Durham, North Carolina
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Pittsburgh, Pennsylvania
  - Study Site, Nashville, Tennessee
  - Study Site, Houston, Texas
  - Study Site, Richmond, Virginia

REFERENCES:
- [Result] Ataga KI, Smith WR, De Castro LM, Swerdlow P, Saunthararajah Y, Castro O, Vichinsky E, Kutlar A, Orringer EP, Rigdon GC, Stocker JW; ICA-17043-05 Investigators. Efficacy and safety of the Gardos channel blocker, senicapoc (ICA-17043), in patients with sickle cell anemia. Blood. 2008 Apr 15;111(8):3991-7. doi: 10.1182/blood-2007-08-110098. Epub 2008 Jan 11. PMID 18192510
- See also: For more information about Icagen — http://www.icagen.com
- See also: For more information about Sickle Cell Disease — http://www.SCInfo.org